CLINICAL TRIAL: NCT03999372
Title: Evaluation of Sperm Selection Technique Using Hyaluronic Acid Binding in Intra-cytoplasmic Sperm Injection (ICSI)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ClinAmygate (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Clin-I-0201909
Record Dates: First submitted 2019-06-25; First posted 2019-06-26 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Infertility, Male
MeSH Terms: conditions — Infertility, Male | interventions — Sperm Injections, Intracytoplasmic

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: neither the participant nor the outcomes assessor know the assignment codes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PICSI procedure (Experimental): PICSI procedure: PICSI dishes are conventional plastic culture dishes pre-prepared with 3 microdots of powdered. The powdered HA is re-hydrated by adding 5 μL droplets of fresh culture medium to each of the three microdots. A 2 μL droplet with suspension of treated spermatozoa is then connected with a pipette tip to these culture medium droplets. The PICSI dish is incubated under oil; within 5 minutes the bound spermatozoa are attached by their head to the surface of the HA-microdots and are spinning around their head. An ICSI injecting pipette is used to pick the best motile HA-bound sperm up and inject them one by one into an oocyte. The ICSI injecting pipette can be previously loaded with viscous medium (PVP or Sperm Slow) to facilitate sperm micromanipulation.
  Interventions: Biological: Hyaluronan binding system
- ICSI procedure (Active Comparator): ICSI procedure: following sperm preparation as described before, samples were incubated until time of injection. Each oocyte was injected with a single morphologically abnormal and immobilized in polyvinyl Pyrolidone (PVP) spermatozoon. Individual sperm subjected to ICSI was examined and evaluated. The injection procedure was carried out in a sterilized dish using holding pipette and injection needle. Intra cytoplasmic sperm injection was performed according to the protocol of Van Steirteghem.
  Interventions: Other: ICSI

INTERVENTIONS:
Biological: Hyaluronan binding system — Hyaluronan binding system for sperm selection for ICSI procedures (PICSI)
  Arms: PICSI procedure
Other: ICSI — Normal ICSI procedure
  Arms: ICSI procedure

SUMMARY:
In vitro sperm selection for ICSI is important as it has a direct influence on the paternal contribution of preimplantation embryogenesis. Various laboratory tests were developed to assess the functions of the spermatozoa. Among them, only the tests for sperm DNA fragmentation, hyperactivation of the spermatozoa and the hyaluronan-binding ability are simple and fast.

DETAILED DESCRIPTION:
In vitro sperm selection for ICSI is important as it has a direct influence on the paternal contribution of preimplantation embryogenesis. Men with oligozoospermia who require ICSI often demonstrate compromised DNA integrity and increased chromosomal aberrations of the sperms in their semen. Studies have shown that embryos resulting from ICSI in those men have higher risk of sex chromosome disomies, chromosomal aneuploidies, de novo numerical chromosomal aberrations and cytogenetically detectable structural chromosomal aberrations. Although the main candidates for ICSI are oligozoospermic men, there is an increase in the use of ICSI, therefore, more couples are potentially exposed to those potential risks.

Various laboratory tests were developed to assess the functions of the spermatozoa. Among them, only the tests for sperm DNA fragmentation (Halosperm), hyperactivation of the spermatozoa and the hyaluronan-binding ability (HBA) are simple and fast enough to allow the same semen sample tested to be used for oocytes' insemination. Spermatozoa that are fail to bind to hyaluronan have many aspects of immaturity. They retain histones in the sperm nucleus, cytoplasm on the sperm neck, and have higher aberrant sperm head morphology, in addition to, lower genomic integrity. It has also been shown that sperm DNA fragmentation is associated with male factor of infertility, correlating with the morphology and motility of spermatozoa.

The aim of the present study is to carry out a comparative analysis between two groups: Hyaluronan binding system for sperm selection for ICSI procedures and another group of conventional morphology sperm selection (ICSI-PVP), both in cycles with only male infertility factor. The evaluated parameters were semen quality, fertilization and cleavage rates, chemical and clinical pregnancy, and miscarriage rates.

ELIGIBILITY:
Inclusion Criteria:

* Female 20-40 years
* Male factor infertility

Exclusion Criteria:

* Other factor of infertility (tubal, uterine, ... etc)

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 300 (Actual)
Dates: Start 2019-07-05 (Actual); Primary Completion 2019-12-02 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | Up to 2 weeks
  Clinical pregnancy rate (viable fetus)

SECONDARY OUTCOMES:
Number of high quality embryos | Within 48 hours of fertilization
  Number of high quality embryos

CONTACTS AND LOCATIONS:
Overall Officials: Eman Elgendy, MD, Principal Investigator — International Islamic Centre for Population Studies and Research
Locations (2):
- Egypt (2):
  - Alazahr University, Cairo
  - Assisted Reproduction Unit International Islamic Centre for Population Studies and Research, Al-Azhar University, Cairo

IPD SHARING:
Plan to Share IPD: No
As per our local regulations

REFERENCES:
- [Background] Worrilow KC, Eid S, Woodhouse D, Perloe M, Smith S, Witmyer J, Ivani K, Khoury C, Ball GD, Elliot T, Lieberman J. Use of hyaluronan in the selection of sperm for intracytoplasmic sperm injection (ICSI): significant improvement in clinical outcomes--multicenter, double-blinded and randomized controlled trial. Hum Reprod. 2013 Feb;28(2):306-14. doi: 10.1093/humrep/des417. Epub 2012 Nov 30. PMID 23203216